CLINICAL TRIAL: NCT04478019
Title: Role of NaSo-oropHaryngeal Antiseptic dEcolonizaiton to Reduce Covid-19 Viral Shedding and Disease Transmission: SHIELD Study
Brief Title: SHIELD Study: Using Naso-oropharyngeal Antiseptic Decolonization to Reduce COVID-19 Viral Shedding
Acronym: SHIELD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0540; A534265 (Other: UW Madison); SMPH/MEDICINE/INFECT DIS (Other: UW Madison); Protocol Version 6/1/2020 (Other: UW Madison)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; SARS-CoV 2
Keywords: COVID-19; povidone-iodine; chlorhexidine gluconate; transmission; virology
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Two-period cross-over trial with a wash-out period between two study intervention periods. Participants will be randomized in a 1:1 ratio to two intervention sequences: active intervention followed by a no intervention control; or no intervention control followed by active intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control > Active Intervention (Other): Treatment is 3 weeks of standard personal protective equipment without any povidone-iodine (PI) or chlorhexidine gluconate (CHG) intervention (control), followed by a 2 weeks washout period, and 3 weeks of nasal (10% povidone-iodine swab sticks in each nostril) and CHG oral decolonization (swish and spit 15 ml 0.12% CHG oral rinse for 30 seconds, four times/day) procedures.
  Interventions: Drug: 10% Povidone-iodine nasal decolonization swab plus 0.12% CHG oral rinse
- Active Intervention > Control (Other): Treatment is 3 weeks of nasal (10% povidone-iodine swab sticks in each nostril) and CHG oral decolonization (swish and spit 15 ml 0.12% CHG oral rinse for 30 seconds, four times/day) procedures, followed by 2 weeks of washout, and 3 weeks of standard personal protective equipment without any PI or CHG intervention (control).
  Interventions: Drug: 10% Povidone-iodine nasal decolonization swab plus 0.12% CHG oral rinse

INTERVENTIONS:
Drug: 10% Povidone-iodine nasal decolonization swab plus 0.12% CHG oral rinse — 2 swab sticks of 10% povidone-iodine in each nares and 0.12% CHG oral rinse

SUMMARY:
Essential workers in positions with increased likelihood of exposure to SARS-CoC-2 will be most impacted by the proposed project. Evidence has shown that the SARS-CoV-2 novel coronavirus is easily transmissable through close contact between individuals, especially during aerosol-generating procedures such as intubation of patients. The intervention proposed in this study (nasal and oral decontamination with povidone-iodine and chlorhexidine, respectively) presents an opportunity for a safe, effective, and feasible treatment to decontaminate the primary entry points for SARS-CoV-2. As such, the intervention to be studied in this project may protect healthcare and other essential workers by preventing transmission of SARS-CoV-2 from patients to healthcare workers, as well as the general public to essential worker,. and thus reducing the incidence of COVID-19 in these workers.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a essential worker performing at least some in-person job duties (not 100% remote)
* Participant is willing and able to perform intervention and data collection procedures.
* Participant is able to provide informed consent in English language.

Exclusion Criteria:

* Diagnosis of COVID-19 within 2 months prior to enrollment, or active respiratory illness symptoms at time of enrollment
* Known medical contraindication to chlorhexidine gluconate or povidone-iodine treatment ingredients (such as a known allergy)
* Participant has a known medical and/or surgical reason prohibiting nasal swab sampling.
* Participant is female who is pregnant, or believes she may be pregnant, at time of enrollment.
* Participant is actively taking/using any treatments or interventions as part of any other COVID-19 related investigational trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with COVID-19 diagnosis | 8 weeks
  Participants will be monitored for positive COVID-19 test results during this trial
SARS-Cov-2 Viral Load | 8 weeks
  Viral load will be measured as a continuous outcome for each participant (three times per week) throughout this trial.

SECONDARY OUTCOMES:
Fidelity of the treatment regimen | 8 weeks
  Assessment of fidelity (as measured by percentage of compliance) to the treatment regimen will be measured by participants' reporting of intervention doses take through a daily treatment diary.
Feasibility of the treatment regimen | 2 weeks total: 1 week (pre-intervention) and 1 week after completion of intervention (post-intervention)
  A survey asking subjects to rank several factors that contribute to overall feasibility of use will be given pre- and post-intervention treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study results will be shared with other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared after enrollment goals are reached for this study. Data will be shared via this website and publication in peer-reviewed journals.